CLINICAL TRIAL: NCT05481216
Title: HIV-1 & Coronavirus-Coinfection in Europe: Morbidity & Risk Factors of COVID-19 in People Living With HIV
Acronym: HIV CoCo
Status: Completed | Type: Observational
Sponsor: NEAT ID Foundation (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 303CoCo
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: HIV-1-infection; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PLWHIV with COVID-19 cases: Patients who are at least 18 years of age with documented HIV-1 infection and confirmed SARS-CoV-2 infection by documented, or patient-reported, positive result on PCR testing of a nasopharyngeal or respiratory sample, before 1st April 2021.
  Interventions: Other: COVID-19; Other: HIV-1 infection
- PLWHIV without COVID-19 controls: Patients at least 18 years of age with documented HIV-1 infection.
  Interventions: Other: HIV-1 infection
- HIV seronegative patients with COVID-19 controls: Patients at least 18 years of age with confirmed SARS-CoV-2 infection by documented, or patient-reported, positive result on PCR testing of a nasopharyngeal or respiratory sample, before 1st April 2021.
  Interventions: Other: COVID-19

INTERVENTIONS:
Other: COVID-19 — Diagnosed with COVID-19 infection
  Groups: HIV seronegative patients with COVID-19 controls; PLWHIV with COVID-19 cases
Other: HIV-1 infection — Diagnosed with HIV-1 infection
  Groups: PLWHIV with COVID-19 cases; PLWHIV without COVID-19 controls

SUMMARY:
HIV CoCo is a European multi-centre, multi-country, retrospective, observational case-control study that will aim to describe clinical outcomes and identify risk factors for People Living With HIV (PLWHIV) who are co-infected with the SARS-CoV-2 coronavirus.

The study will address two central questions:

1. Is there a particular risk for COVID-19 in PLWHIV as compared to HIV seronegative control COVID-19 cases?
2. Are there particular factors, within the group of PLWHIV, which put them at risk for a more severe COVID-19 disease course?

The study will address these questions by recruiting patients co-infected with both HIV and SARS-CoV-2 and comparing them to two control groups - one group infected with SARS-CoV-2 only and another group infected with HIV only. Only deidentified, real-world retrospective data will be used for the study, collected as part of standard, routine clinical care.

Additionally, this study will also look to:

1. Describe the differences in the clinical manifestation of COVID-19 in PLWHIV compared to HIV seronegative controls
2. Describe the response to treatment, including supportive care and novel therapies against COVID-19, including antiviral or immunomodulatory therapy
3. Describe the co-morbidities in PLWHIV and controls with COVID-19
4. Compare the severity of COVID-19 between PLWHIV and the COVID-19 only controls at diagnosis and hospital admission.

Data will be collected about patient outcomes from COVID-19 (including hospitalisation for COVID-19, length of stay in hospital, critical care admission, ventilation/oxygenation requirements, and need for kidney replacement therapy), as well as pre-existing health conditions, and relevant blood results at COVID-19 diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* • Cases (PLWHIV + COVID-19)

  1. Any gender
  2. At least 18 years of age
  3. Documented HIV-1 infection
  4. Confirmed SARS-CoV-2 infection by documented, or patient-reported, positive result on PCR testing of a nasopharyngeal or respiratory sample, before 1st April 2021

     * Controls (COVID-19)

  <!-- -->

  1. Any gender
  2. At least 18 years of age
  3. No documented HIV-1 infection
  4. Confirmed SARS-CoV-2 infection by documented, or patient-reported, positive result on PCR testing of a nasopharyngeal or respiratory sample, before 1st April 2021
  5. Meet the matching criteria

For comparing PLWHIV & COVID-19 versus HIV seronegative COVID-19 patients, a 1:1 matching will be performed according to the following criteria:

* Age (+/- 5 years)
* Sex
* Ethnicity (where available)
* Month of COVID-19 diagnosis (+/- 2 months)
* COVID-19 diagnosis inpatient OR
* COVID-19 diagnosis outpatient (ambulatory)
* Controls (PLWHIV)

  1. Any gender
  2. At least 18 years of age
  3. Documented HIV-1 infection
  4. No evidence of SARS-CoV-2 infection
  5. Meet the matching criteria

For comparing PLWHIV & COVID-19 versus PLWHIV without COVID-19, a 1:2 matching for similar risk of acquiring COVID-19 will be performed according to the following criteria:

* Age (+/- 5 years)
* Sex
* Ethnicity (where available)

Exclusion Criteria

For cases (PLWHIV + COVID-19) and for COVID-19 only controls:

* COVID-19 diagnosed based on clinical criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult PLWHIV with and without COVID-19 disease, followed up at the study sites for routine clinical care. Data from adult COVID-19 patients without HIV infection will be used as controls.
  500 cases (PLWHIV + COVID-19) will be recruited. These patients will be at least 18 years old with documented HIV-1 infection and SARS-CoV-2 infection by documented, or patient-reported, positive result on PCR testing of a nasopharyngeal or respiratory sample, before 1st April 2021.
  500 COVID-19 controls will be recruited. These patients will be at least 18 years old without documented HIV-1 infection but confirmed SARS-CoV-2 infection by documented, or patient-reported, positive result on PCR testing of a nasopharyngeal or respiratory sample, before 1st April 2021.
  1000 PLWHIV control patients will be recruited for the second control group. This group will include individuals at least 18 years old with documented HIV-1 infection.
Sampling Method: Non-Probability Sample
Enrollment: 2598 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- CHU Saint Pierre, Brussels, Belgium
- France (2):
  - Hôpital Européen Marseille, Marseille
  - Hôpital Saint Louis, Paris
- Erasmus Medical Center, Rotterdam, Netherlands
- Spain (10):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario San Pedro, Logroño
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
- United Kingdom (9):
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Southmead Hospital (North Bristol), Bristol
  - University Hospitals of Derby & Burton NHS Foundation Trust, Derby
  - Brownlee Centre, Gartnavel General Hospital, Glasgow
  - Barts Health (The Royal London Hospital), London
  - Chelsea & Westminster Hospital NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Only anonymised summary-format data will be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PLWH were identified from European sites in the NEAT ID network. PLWH are routinely followed-up at specialized outpatient clinics with regular follow up visits as standard of care. HIV-COVID+ inpatient controls were from the same sites of the NEAT ID network. HIV-COVID-19+ outpatient controls were from the anonymized real-world primary care medical database THIN.
Pre-assignment Details: PCR-confirmed SARS-CoV-2 infected PLWH (HIV+COVID+) were matched 1:1(outpatient) or 1:3(inpatient )against HIV negative PCR-confirmed COVID-19-infected individuals (HIV-COVID+) and 1:2 COVID-19 negative PLWH (HIV+COVID-).
Period: Overall Study
Arm/Group | PLWHIV With COVID-19 Cases | PLWHIV Without COVID-19 Controls | HIV Seronegative Patients With COVID-19 Controls
Started | 500 | 992 | 1106
Completed | 500 | 992 | 1106
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 486 HIV+COVID+ cases were included in the analysis of HIV+COVID+ vs HIV-COVID+ (14 cases lacked COVID+ inpatient controls).Co-morbidities were only available for 395 cases except for peripheral vascular disease, dementia and hemiplegia which were available for 320 cases. The case and control groups do not come from the same population and could not be grouped together for all baseline characteristics. Total population data that could be calculated from the data collected has been reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLWHIV With COVID-19 Cases | PLWHIV Without COVID-19 Controls | HIV Seronegative Patients With COVID-19 Controls | Total
Number analyzed (Participants) | 500 | 992 | 1106 | 2598
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11.3) | 52 (11.1) | 51 (11.1) | 51.6 (11.2)
Age, Customized [Count of Participants; unit: Participants]
  Age (years): <60 years | 388 | 778 | 878 | 2044
  Age (years): ≥ 60 years | 112 | 214 | 228 | 554
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 348 | 409 | 933
  Male | 324 | 644 | 697 | 1665
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Ethnicity was not available for 762 HIV-COVID-19+ outpatient control cases obtained from the anonymized real-world primary care medical database THIN.
  Participants
    Ethnicity: number analyzed (Participants) | 500 | 992 | 344 | 1836
    Ethnicity: White Caucasian | 226 | 464 | 148 | 838
    Ethnicity: White Mixed | 37 | 49 | 24 | 110
    Ethnicity: Asian | 4 | 7 | 4 | 15
    Ethnicity: Black | 163 | 329 | 86 | 578
    Ethnicity: Other | 12 | 23 | 4 | 39
    Ethnicity: Not stated | 58 | 120 | 78 | 256
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 38 | 24 | 78 | 140
  Belgium | 50 | 4 | 144 | 198
  United Kingdom | 194 | 166 | 333 | 693
  France | 53 | 682 | 230 | 965
  Spain | 165 | 116 | 321 | 602
Month of COVID-19 diagnosis [Median (Inter-Quartile Range); unit: month/year] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. 486 HIV+COVID+ cases were included in the HIV+COVID+ vs HIV-COVID+ analysis because 14 cases lacked HIV-COVID+ inpatient controls and were excluded.
  month/year
    number analyzed (Participants) | 486 | 0 | 1106 | 1592
    (all) | 102020 [042020 to 122020] |  | 102020 [042020 to 122020] | 102020 [042020 to 122020]
COVID-19 diagnosis location [Number; unit: Diagnosis location] — Population: 486 HIV+COVID+ vs HIV-COVID+ included in the analysis because 14 cases lacked COVID+ inpatient controls.
  Diagnosis location
    Inpatient: number analyzed (Participants) | 486 | 0 | 1106 | 1592
    Inpatient | 176 |  | 176 | 352
    Outpatient: number analyzed (Participants) | 486 | 0 | 1106 | 1592
    Outpatient | 310 |  | 930 | 1240
Body weight [Mean (Standard Deviation); unit: kg] — Population: Due to the retrospective nature of this data collection study, data collection was limited to available data. Baseline weight characteristics were available for 479 HIV+COVID-19+ cases, 779 HIV-COVID+ controls and 943 HIV+COVID- controls
  kg
    number analyzed (Participants) | 479 | 943 | 779 | 2201
    (all) | 82 (17.1) | 79 (16.1) | 81 (19.1) | 80.4 (17.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Due to the retrospective nature of this data collection study, data collection was limited to available data. Baseline body mass index data only available for 428 COVID-19+HIV+ cases, 847 COVID-19- HIV+ and 581 COVID-19+HIV- controls.
  kg/m^2
    number analyzed (Participants) | 428 | 847 | 581 | 1856
    (all) | 28.1 (6.0) | 26.8 (5.4) | 28.7 (6.2) | 27.7 (5.9)
Comorbidities [Count of Participants; unit: Participants] — Population: Due to the retrospective nature of this data collection study, data collection was limited to available data. Baseline comorbidity data was only available for 634 HIV-COVID+ controls except for peripheral vascular disease, dementia and hemiplegia which was only available for 344 controls.
  Participants
    Myocardial Infarction: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Myocardial Infarction | 16 | 34 | 17 | 67
    Congestive Heart Failure: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Congestive Heart Failure | 13 | 20 | 21 | 54
    Peripheral Vascular Disease: number analyzed (Participants) | 500 | 992 | 344 | 1836
    Peripheral Vascular Disease | 28 | 42 | 9 | 79
    Cerebrovascular Accident: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Cerebrovascular Accident | 19 | 25 | 24 | 68
    Dementia: number analyzed (Participants) | 500 | 992 | 344 | 1836
    Dementia | 16 | 19 | 6 | 41
    Chronic Obstructive Pulmonary Disease: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Chronic Obstructive Pulmonary Disease | 36 | 43 | 35 | 114
    History of Pneumonia: number analyzed (Participants) | 500 | 992 | 634 | 2126
    History of Pneumonia | 83 | 146 | 46 | 275
    Connective Tissue Disease: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Connective Tissue Disease | 21 | 25 | 144 | 190
    Peptic Ulcer Disease: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Peptic Ulcer Disease | 21 | 35 | 30 | 86
    Liver Disease: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Liver Disease | 69 | 141 | 54 | 264
    Diabetes: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Diabetes | 59 | 97 | 131 | 287
    Hemiplegia: number analyzed (Participants) | 500 | 992 | 344 | 1836
    Hemiplegia | 2 | 3 | 0 | 5
    Paralysis of Arm(s) or Leg(s): number analyzed (Participants) | 500 | 992 | 634 | 2126
    Paralysis of Arm(s) or Leg(s) | 3 | 3 | 6 | 12
    Chronic Kidney Disease: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Chronic Kidney Disease | 38 | 32 | 14 | 84
    Current or history of Cancer: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Current or history of Cancer | 46 | 99 | 79 | 224
    Leukemia: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Leukemia | 1 | 3 | 3 | 7
    Lymphoma: number analyzed (Participants) | 500 | 992 | 634 | 2126
    Lymphoma | 12 | 30 | 10 | 52
Drug treatment for COVID-19 [Count of Participants; unit: Participants] — Population: Drug treatment data was not available for the overall population
  Participants
    Glucocorticoids: number analyzed (Participants) | 109 | 0 | 109 | 218
    Glucocorticoids | 32 |  | 53 | 85
    Azithromycin: number analyzed (Participants) | 109 | 0 | 109 | 218
    Azithromycin | 39 |  | 46 | 85
    Other antibiotics: number analyzed (Participants) | 109 | 0 | 109 | 218
    Other antibiotics | 39 |  | 44 | 83
    Hydroxychloroquine: number analyzed (Participants) | 126 | 0 | 129 | 255
    Hydroxychloroquine | 62 |  | 49 | 111
    Remdesivir: number analyzed (Participants) | 126 | 0 | 129 | 255
    Remdesivir | 9 |  | 14 | 23
    Tocilizumab: number analyzed (Participants) | 126 | 0 | 129 | 255
    Tocilizumab | 5 |  | 3 | 8
    Monoclonal antibodies against SARS-CoV2: number analyzed (Participants) | 126 | 0 | 129 | 255
    Monoclonal antibodies against SARS-CoV2 | 1 |  | 7 | 8
    Reconvalescent plasma: number analyzed (Participants) | 126 | 0 | 129 | 255
    Reconvalescent plasma | 3 |  | 1 | 4
    Anti-IL1 Inhibitors: number analyzed (Participants) | 126 | 0 | 129 | 255
    Anti-IL1 Inhibitors | 2 |  | 1 | 3
    Anti-IL6 Inhibitors: number analyzed (Participants) | 126 | 0 | 129 | 255
    Anti-IL6 Inhibitors | 8 |  | 20 | 28
    Lopinavir/ritonavir: number analyzed (Participants) | 126 | 0 | 129 | 255
    Lopinavir/ritonavir | 25 |  | 36 | 61
    Anticoagulants: number analyzed (Participants) | 109 | 0 | 109 | 218
    Anticoagulants | 13 |  | 18 | 31
    Others: number analyzed (Participants) | 109 | 0 | 109 | 218
    Others | 18 |  | 33 | 51
Blood cell counts at COVID-19 diagnosis [Mean (Standard Deviation); unit: 10^9/L cells] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the retrospective nature of this data collection study, data collection was limited to available data. Blood cell counts were not available for all participants
  10^9/L cells
    Platelet count: number analyzed (Participants) | 180 | 0 | 185 | 365
    Platelet count | 212 (87.9) |  | 237 (105.5) | 225 (97.9)
    WBC count: number analyzed (Participants) | 178 | 0 | 183 | 361
    WBC count | 7.2 (3.5) |  | 7.4 (4.1) | 7.3 (3.8)
    Neutrophils: number analyzed (Participants) | 165 | 0 | 169 | 334
    Neutrophils | 7.0 (11.9) |  | 8.3 (14.3) | 7.7 (13.2)
    Lymphocytes: number analyzed (Participants) | 168 | 0 | 171 | 339
    Lymphocytes | 2.0 (3.9) |  | 1.8 (3.2) | 1.9 (3.6)
    Monocytes: number analyzed (Participants) | 167 | 0 | 170 | 337
    Monocytes | 1.0 (3.3) |  | 0.7 (1.1) | 0.8 (2.5)
    Eosinophils: number analyzed (Participants) | 162 | 0 | 166 | 328
    Eosinophils | 0.07 (0.12) |  | 0.13 (0.59) | 0.10 (0.42)
    Basophils: number analyzed (Participants) | 160 | 0 | 163 | 323
    Basophils | 0.05 (0.17) |  | 0.04 (0.16) | 0.05 (0.16)
Inflammatory Markers and Kidney Function Tests [Mean (Standard Deviation); unit: mg/dL] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection study, data collection was limited to available data. Inflammatory Markers and Kidney Function Tests were not available for all participants and could not be collected.
  mg/dL
    Total bilirubin: number analyzed (Participants) | 151 | 0 | 152 | 303
    Total bilirubin | 0.7 (0.9) |  | 0.7 (0.9) | 0.7 (0.9)
    Urea: number analyzed (Participants) | 144 | 0 | 145 | 289
    Urea | 52.6 (64.0) |  | 39.7 (30.2) | 46.1 (50.3)
    Serum creatinine: number analyzed (Participants) | 173 | 0 | 176 | 349
    Serum creatinine | 1.8 (3.3) |  | 1.1 (1.1) | 1.4 (2.5)
    Calcium: number analyzed (Participants) | 96 | 0 | 96 | 192
    Calcium | 4.9 (3.2) |  | 5.7 (9.0) | 5.3 (6.7)
RBC Count at COVID-19 Diagnosis [Mean (Standard Deviation); unit: 10^12/L cells] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection study, data collection was limited to available data. Blood cell counts were not available for all participants and could not be collected
  10^12/L cells
    number analyzed (Participants) | 172 | 0 | 177 | 349
    (all) | 4.4 (0.8) |  | 4.6 (0.7) | 4.5 (0.8)
Haemoglobin at COVID-19 diagnosis [Mean (Standard Deviation); unit: g/dL] — Population: This measure is only applicable to COVID+ participants and was not collected for HIV+COVID- controls. As this is a real world retrospective data collection study, there are limitations in data availability and Haemoglobin values were not available for all participants. Data was available for 178 HIV+COVID+ cases and 183 HIV-COVID+ controls.
  g/dL
    number analyzed (Participants) | 178 | 0 | 183 | 361
    (all) | 13.0 (2.3) |  | 13.1 (2.2) | 13.1 (2.2)
Haematocrit at COVID-19 diagnosis [Mean (Standard Deviation); unit: L/L] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection study, data collection was limited to available data. Haematocrit not available for all participants in the analysis population
  L/L
    number analyzed (Participants) | 173 | 0 | 178 | 351
    (all) | 2.8 (3.0) |  | 2.8 (3.3) | 2.8 (3.2)
Glucose, Cholesterol and Triglycerides at COVID-19 diagnosis [Mean (Standard Deviation); unit: mmol/L] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection study, data collection was limited to available data. Data was not available for all participants in the analysis population
  mmol/L
    Glucose: number analyzed (Participants) | 94 | 0 | 98 | 192
    Glucose | 7.0 (3.6) |  | 7.4 (5.1) | 7.2 (4.4)
    Total cholesterol: number analyzed (Participants) | 31 | 0 | 31 | 62
    Total cholesterol | 4.4 (0.9) |  | 3.8 (1.3) | 4.1 (1.1)
    Triglycerides: number analyzed (Participants) | 34 | 0 | 34 | 68
    Triglycerides | 1.6 (0.9) |  | 1.9 (1.3) | 1.8 (1.1)
MCV at COVID diagnosis [Mean (Standard Deviation); unit: fL] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection study, data collection was limited to available data. Data was not available for all participants in the analysis population
  fL
    number analyzed (Participants) | 176 | 0 | 181 | 357
    (all) | 91.4 (7.3) |  | 87.3 (8.6) | 89.3 (8.2)
MCH at COVID-19 diagnosis [Mean (Standard Deviation); unit: pg] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection study, data collection was limited to available data. Data was not available for all participants in the analysis population
  pg
    number analyzed (Participants) | 171 | 0 | 175 | 346
    (all) | 30.2 (2.8) |  | 29.1 (2.4) | 29.6 (2.7)
Lactate dehydrogenase, ALT and AST levels at COVID-19 diagnosis [Mean (Standard Deviation); unit: U/L] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection study, data collection was limited to available data. Data not available for all participants in the analysis population
  U/L
    ALT: number analyzed (Participants) | 156 | 0 | 158 | 314
    ALT | 42.0 (78.9) |  | 47.4 (44.7) | 44.7 (63.9)
    AST: number analyzed (Participants) | 122 | 0 | 124 | 246
    AST | 55.2 (118.4) |  | 54.0 (50.5) | 54.6 (90.6)
    Lactate dehydrogenase: number analyzed (Participants) | 86 | 0 | 86 | 172
    Lactate dehydrogenase | 357.5 (205.3) |  | 412.2 (237.1) | 384.9 (222.8)
HbA1C levels at COVID-19 diagnosis [Mean (Standard Deviation); unit: mmol/mol] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection study, data collection was limited to available data. Data was not available for all participants in the analysis population
  mmol/mol
    number analyzed (Participants) | 4 | 0 | 4 | 8
    (all) | 60.5 (36.7) |  | 99.9 (72.0) | 79.9 (56.8)
C-Reactive Protein (CRP) at COVID-19 diagnosis [Mean (Standard Deviation); unit: mg/L] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection, data collection was limited to available data. CRP levels were not available for all participants and could not be collected
  mg/L
    number analyzed (Participants) | 129 | 0 | 131 | 260
    (all) | 12.6 (18.7) |  | 13.6 (21.8) | 13.1 (20.3)
Ferritin and D-dimer levels at COVID-19 diagnosis [Mean (Standard Deviation); unit: ng/mL] — Population: This measure is only applicable to the HIV-COVID+ and HIV+COVID+ populations. Due to the nature of this retrospective data collection, data collection was limited to available data. Ferritin levels and D-dimer were not available for all participants and could not be analysed.
  ng/mL
    Ferritin: number analyzed (Participants) | 58 | 0 | 59 | 117
    Ferritin | 1039.5 (1398.8) |  | 1113.0 (1143.6) | 1076.6 (1271.5)
    D-dimer: number analyzed (Participants) | 87 | 0 | 87 | 174
    D-dimer | 1653.8 (2452.7) |  | 1561.9 (2299.8) | 1607.9 (2371.0)
Time since HIV diagnosis [Mean (Standard Deviation); unit: years] — Population: This measure not applicable to HIV seronegative population. Due to the nature of this retrospective data collection study, data collection was limited to available data. Data was not available for all participants and could not be analysed.
  years
    number analyzed (Participants) | 492 | 977 | 0 | 1469
    (all) | 17.8 (9.5) | 18.7 (9.3) |  | 18.4 (9.4)
CD4 cell count [Mean (Standard Deviation); unit: cells/mm^3] — Population: This measure not applicable to HIV seronegative population. Due to the nature of this retrospective data collection study, data collection was limited to available data. CD4 count was not available for all participants and could not be analysed.
  cells/mm^3
    number analyzed (Participants) | 489 | 971 | 0 | 1460
    (all) | 654 (332.9) | 669 (321.9) |  | 664 (325.6)
HIV viral load [Count of Participants; unit: Participants] — Population: This measure not applicable to HIV seronegative population. Due to the nature of this retrospective data collection study, data collection was limited to available data. HIV viral load was not available for all participants and could not be analysed.
  Participants
    <50 copies/ml: number analyzed (Participants) | 492 | 976 | 0 | 1468
    <50 copies/ml | 423 | 878 |  | 1301
    ≥50 copies/ml: number analyzed (Participants) | 492 | 976 | 0 | 1468
    ≥50 copies/ml | 69 | 98 |  | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Composite Primary End Point (Critical Care Admission, Palliative Discharge When Discharged From Hospital, or Mortality Within the 6 Weeks After Diagnosis of COVID-19) Events
Description: The primary endpoint is a composite of the number of critical care admission (high dependency unit or intensive care unit), mortality in hospital or palliative discharge when discharged from hospital, or mortality at 6 weeks after diagnosis of COVID-19 or at discharge from hospital (where applicable) events. Time-to-event methods, including Kaplan-Meier survival curves and Cox proportional-hazards models, will be used for this analysis. The time to the primary endpoints will be defined as:
  * For participants admitted to critical care Time = [Date of Critical care admission - Date of positive PCR test for COVID-19] + 1
  * For participants admitted to critical care before diagnosis of COVID-19, Time=1 day.
  * For participants with palliative discharge when discharged from hospital Time = [Date of discharge from hospital to palliative care - Date of positive PCR test for COVID-19] + 1.
  * For participants died Time = [Date of death - Date of positive PCR test for COVID-19] + 1.
Time Frame: From baseline (diagnosis of COVID-19) to Week 6
Population: There were 486 HIV+COVID+ cases included in the analysis as 14 cases lacked HIV-COVID+ inpatient controls and were excluded. This outcome was analysed in participants diagnosed with COVID-19 and is not applicable and not reported to the HIV+COVID-19- arm.
Measure: Number; unit: Events
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 486 | 1106
Events | 66 | 67

2. Primary Outcome: Kaplan-Meier Estimate of Primary End Point
Description: Kaplan-Meier estimate of the composite number of critical care admission, palliative discharge and death events
Time Frame: From Baseline (diagnosis of COVID-19 ) to week 6
Population: There were 486 HIV+COVID+ cases included in the analysis as 14 cases lacked HIV-COVID+ inpatient controls and were excluded. This measure was analysed in participants diagnosed with COVID-19 and is not reported for the HIV+COVID-19- arm.
Measure: Number (95% Confidence Interval); unit: percentage of events
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 486 | 1106
percentage of events | 13.6 [10.8 to 17.0] | 6.1 [4.8 to 7.6]
Statistical Analysis 1: Comparison: PLWHIV With COVID-19 Cases vs HIV Seronegative Patients With COVID-19 Controls; Test type: Other — Unadjusted and adjusted hazard ratios (HR) will be calculated using a proportional Cox regression model. The adjusted variables were body mass index (BMI), dementia, peripheral vascular disease, history of pneumonia, connective tissue disease, liver disease, diabetes, chronic kidney disease, glucocorticoids, hydroxychloroquine, tocilizumab, and anti-IL6 inhibitors; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.73 to 2.29]
Statistical Analysis 2: Comparison: PLWHIV With COVID-19 Cases vs HIV Seronegative Patients With COVID-19 Controls; The adjusted variables were body mass index (BMI), dementia, peripheral vascular disease, history of pneumonia, connective tissue disease, liver disease, diabetes, chronic kidney disease, glucocorticoids, hydroxychloroquine, tocilizumab, and anti-IL6 inhibitors; Test type: Other; Adjusted Hazard Ratio = 1.30, 95% CI 2-sided [0.73 to 2.29]

3. Primary Outcome: Number of Palliative Discharge
Description: Number of palliative discharge at discharge from hospital following hospitalisation for COVID-19 events
Time Frame: Baseline (diagnosis of COVID-19) to week 6
Population: 486 HIV+COVID+ vs HIV-COVID+ were included in the analysis as 14 HIV+COVID+ cases lacked COVID+ inpatient controls. This measure was analysed for participants with COVID-19 .It is not applicable for COVID-19- participants and not reported for the HIV+COVID-19- arm.
Measure: Count of Participants; unit: Participants
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 486 | 1106
Participants | 1 | 0

4. Primary Outcome: Mortality
Description: Mortality at 6 weeks after diagnosis of COVID-19 or at discharge from hospital
Time Frame: Baseline (diagnosis of COVID-19) to week 6
Population: 486 HIV+COVID+ vs HIV-COVID+ were included in the analysis as 14 HIV+COVID+ cases lacked COVID+ inpatient controls and were excluded. This measure was analysed for participants with COVID-19. It is not applicable for COVID-19- participants and not reported for the HIV+COVID-19- arm.
Measure: Count of Participants; unit: Participants
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 486 | 1106
Participants | 24 | 23

5. Primary Outcome: Number of Critical Care Admission Events
Description: Number of admission events to a high dependency unit or intensive care unit
Time Frame: Baseline (diagnosis of COVID-19) to week 6
Population: as for outcome 4
Measure: Number; unit: events
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 486 | 1106
events | 55 | 58

6. Primary Outcome: HIV Viral Load
Description: Identification of risk factors for COVID-19 infection within the group of PLHIV: HIV viral load
Time Frame: Baseline(Last CD4 cell count and HIV-RNA before COVID-19 diagnosis, or most recent for PLHIV without COVID-19)
Population: The analysis population will consist of PLHIV and COVID-19 with matched PLHIV without COVID-19. 1:2 matching for similar risk of acquiring COVID-19 will be performed according to the following criteria: Age (+/- 5 years); Sex; Ethnicity (where available). Because some of the variables studied will have missing values, multiple imputation using Chained Equations approach (MICE) will be used to fill in missing data. Ten imputations (M=10) will be chosen.
Measure: Number; unit: copies/ml
Arm/Group | PLWHIV With COVID-19 Cases | PLWHIV Without COVID-19 Controls
Number analyzed (Participants) | 500 | 992
copies/ml
  <50 | 427 | 888
  ≥50 | 73 | 104
Statistical Analysis 1: Comparison: PLWHIV With COVID-19 Cases vs PLWHIV Without COVID-19 Controls; Conditional logistic regression models accounting for case-control matching will be used to identify risk factors for advanced immunodeficiency associated with COVID-19; Test type: Other; p = 0.009, Regression, Logistic

7. Secondary Outcome: Number of Hospitalisation Events
Description: Number of hospital admission for COVID-19 events
Time Frame: Baseline (diagnosis of COVID-19) to week 6
Population: 486 HIV+COVID+ vs HIV-COVID+ were included in the analysis as 14 HIV+COVID+ cases lacked HIV-COVID+ inpatient controls and were excluded. This measure was analysed for participants hospitalised with COVID-19. It is not applicable for COVID-19- participants and not reported for the HIV+COVID-19- arm.
Measure: Number; unit: events
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 486 | 1106
events | 200 | 208

8. Secondary Outcome: Length of Hospital Stay
Description: Length of stay in hospital following hospitalisation for COVID-19
Time Frame: Baseline (diagnosis of COVID-19) to week 6
Population: 486 HIV+COVID+ were included in the analysis as 14 HIV+COVID+ cases lacked HIV-COVID+ inpatient controls and were excluded. This measure was analysed for participants with COVID-19. It is not applicable for COVID-19- participants and not reported for the HIV+COVID-19- arm.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 486 | 1106
days | 11 [9 to 12] | 9 [8 to 11]

9. Secondary Outcome: Length of Stay in ICU
Description: Median Length of Stay in Intensive Care Unit
Time Frame: Baseline (diagnosis of COVID-19) to week 6
Population: 486 HIV+COVID+ vs HIV-COVID+ were included in the analysis as 14 HIV+COVID+ cases lacked COVID+ inpatient controls. This measure was analysed for participants with COVID-19. It is not applicable for COVID-19- participants and not reported for the HIV+COVID-19- arm.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 486 | 1106
days | 18 [11 to 33] | 7 [4 to 21]

10. Secondary Outcome: Ventilator-free Days (VFDs)
Description: Number of ventilator-free days
Time Frame: 6 weeks after diagnosis of COVID-19
Population: Data was not collected
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Extracorporeal Membrane Oxygenation (ECMO)
Description: Length of extracorporeal membrane oxygenation
Time Frame: Baseline (diagnosis of COVID-19) to week 6
Population: Data was not collected
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Need for Kidney Replacement Therapy
Description: The number of patients requiring kidney replacement therapy
Time Frame: Baseline(diagnosis of COVID-19) to week 6
Population: This measure was analysed for participants with COVID-19. It is not applicable for COVID-19- participants and not reported for the HIV+COVID-19- arm. Kidney replacement data was not available for all participants in the HIV+COVID+ and HIV-COVID+ groups due to the retrospective nature of this study, and was only collected for 129 participants per group.
Measure: Number; unit: participants
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 129 | 129
participants | 13 | 6

13. Secondary Outcome: Measurement of Total Comorbidity Burden
Description: Charlson Comorbidity Index predicts the ten-year mortality for a patient who may have a range of comorbid conditions. Index consists of 19 conditions, each with an assigned weight from 1 to 6 according to the relative risk of dying. The total score is derived by summing up the weights of comorbid conditions presented. Based on the CCI score, the severity of comorbidity was categorized into three grades: mild, with CCI scores of 1-2; moderate, with CCI scores of 3-4; and severe, with CCI scores ≥5. The minimum score value is 0 and maximum is 37. A higher score means a more greater mortality risk.
Time Frame: 6 weeks after diagnosis of COVID-19
Population: This measure was analysed for participants with COVID-19. It is not applicable for COVID-19- participants and not reported for the HIV+COVID-19- arm. Co-morbidity data required to analyse this measure was not available for all participants in the HIV+COVID+ and HIV-COVID+ groups due to the retrospective nature of this study, and was only collected for 170 participants per group.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 170 | 170
score on a scale | 2.35 [1.87 to 2.83] | 0.99 [0.82 to 1.16]

14. Secondary Outcome: Estimate Risk of 30-day Mortality After COVID-19 Infection
Description: Estimate risk of 30-day mortality after COVID-19 infection using pre-COVID health status (estimated using the Veterans Health Administration COVID-19 (VACO) index). The VACO index is expressed as a percentage and calculated based on age, sex, Charlson comorbidity index (CCI), and the presence of myocardial infarction (MI) or peripheral vascular disease (PVD). The index range is from 0.2 to 48.0. A higher score means a greater risk of mortality.
Time Frame: Baseline (diagnosis of COVID-19) to week 6
Population: This measure was analysed for participants with COVID-19. It is not applicable for COVID-19- participants and not reported for the HIV+COVID-19- arm. Data required to analyse this measure was not available for all participants in the HIV+COVID+ and HIV-COVID+ groups due to the retrospective nature of this study, and was only collected for 172 participants per group.
Measure: Median (Inter-Quartile Range); unit: percentage of 30- day mortality risk
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 172 | 172
percentage of 30- day mortality risk | 2.65 [2.00 to 5.03] | 2.00 [2.00 to 3.62]

15. Secondary Outcome: Blood Cell Counts at COVID-19 Diagnosis
Description: The endpoint is the blood cell counts at COVID-19 diagnosis. The analyses will be performed with all PLHIV with COVID-19 and matched HIV-uninfected individual with COVID-19 who have data regarding the blood cell count of interest at COVID-19 diagnosis
Time Frame: Baseline (Diagnosis of COVID-19)
Population: Due to the retrospective nature of this data collection study, not all patients in the PLWHIV with COVID and the HIV seronegative with COVID groups had blood cell counts available and could not be included in the analysis. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group.
Measure: Mean (95% Confidence Interval); unit: 10^9/L cells
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 180 | 185
10^9/L cells
  Platelet count | 212.1 [199.4 to 224.9] | 237.2 [221.9 to 252.5]
  WBC count: number analyzed (Participants) | 178 | 183
  WBC count | 7.2 [6.7 to 7.7] | 7.4 [6.8 to 8.0]
  Neutrophils: number analyzed (Participants) | 165 | 169
  Neutrophils | 7.0 [5.2 to 8.8] | 8.3 [6.2 to 10.5]
  Lymphocytes: number analyzed (Participants) | 168 | 171
  Lymphocytes | 2.0 [1.4 to 2.6] | 1.8 [1.3 to 2.3]
  Monocytes: number analyzed (Participants) | 167 | 170
  Monocytes | 1.0 [0.5 to 1.5] | 0.7 [0.5 to 0.8]
  Eosinophils: number analyzed (Participants) | 162 | 166
  Eosinophils | 0.07 [0.05 to 0.08] | 0.13 [0.04 to 0.22]
  Basophils: number analyzed (Participants) | 160 | 163
  Basophils | 0.05 [0.02 to 0.07] | 0.04 [0.04 to 0.06]

16. Secondary Outcome: Liver Function and Tissue Damage Parameters at COVID-19 Diagnosis
Description: The endpoint is the liver function (ALT, AST) and tissue damage (lactate dehydrogenase) parameters at COVID-19 diagnosis.
Time Frame: Baseline(COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had liver function data available and could not be included in the analysis. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group.
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 156 | 158
U/L
  ALT | 42.0 [29.6 to 54.4] | 47.4 [40.4 to 54.4]
  AST: number analyzed (Participants) | 122 | 124
  AST | 55.2 [34.2 to 76.3] | 54.0 [45.0 to 63.0]
  Lactate dehydrogenase: number analyzed (Participants) | 86 | 86
  Lactate dehydrogenase | 357.5 [313.4 to 401.5] | 412.2 [361.3 to 463.0]

17. Secondary Outcome: Inflammatory Markers and Kidney Function Tests
Description: Inflammatory markers and Kidney Function tests at COVID-19 diagnosis
Time Frame: Baseline (COVID-19 Diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had kidney function and inflammatory marker data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 173 | 176
mg/dL
  Total Bilirubin: number analyzed (Participants) | 151 | 152
  Total Bilirubin | 0.7 [0.5 to 0.8] | 0.7 [0.5 to 0.8]
  Urea: number analyzed (Participants) | 144 | 145
  Urea | 52.6 [42.1 to 63.2] | 39.7 [34.8 to 44.7]
  Serum creatinine | 1.8 [1.3 to 2.3] | 1.1 [0.9 to 1.3]
  Calcium: number analyzed (Participants) | 96 | 96
  Calcium | 4.9 [4.2 to 5.5] | 5.7 [3.9 to 7.5]

18. Secondary Outcome: Biological Parameters at COVID-19 Diagnosis
Description: Biological parameters (D-dimer and Ferritin levels) at COVID-19 diagnosis
Time Frame: Baseline(COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had D-dimer and Ferritin levels data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 87 | 87
ng/mL
  D-dimer | 1653.8 [1131.1 to 2176.6] | 1561.9 [1071.8 to 2052.1]
  Ferritin: number analyzed (Participants) | 60 | 61
  Ferritin | 1039.5 [681.2 to 1397.7] | 1113.0 [820.1 to 1405.9]

19. Secondary Outcome: Cholesterol, Triglyceride and Glucose Levels
Description: Cholesterol, Triglyceride and Glucose levels at COVID-19 diagnosis
Time Frame: Baseline(COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had Cholesterol, Triglyceride and Glucose data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 94 | 98
mmol/L
  Total Cholesterol: number analyzed (Participants) | 31 | 31
  Total Cholesterol | 4.4 [4.0 to 4.7] | 3.8 [3.3 to 4.3]
  Total Triglycerides: number analyzed (Participants) | 34 | 34
  Total Triglycerides | 1.6 [1.3 to 1.9] | 1.9 [1.4 to 2.3]
  Glucose | 7.0 [6.3 to 7.7] | 7.4 [6.4 to 8.5]

20. Secondary Outcome: Red Blood Cell Count
Description: Red blood cell (RBC) count at COVID-19 Diagnosis
Time Frame: Baseline(COVID-19 Diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had Red Blood Cell count data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: 10^12/L cells
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 172 | 177
10^12/L cells | 4.4 [4.3 to 4.5] | 4.6 [4.5 to 4.7]

21. Secondary Outcome: Haemoglobin Levels
Description: Haemoglobin levels at COVID-19 diagnosis
Time Frame: Baseline(COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had Haemoglobin data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 178 | 183
g/dL | 13.0 [12.6 to 13.3] | 13.1 [12.8 to 13.5]

22. Secondary Outcome: Haematocrit
Description: Haematocrit levels at COVID-19 diagnosis
Time Frame: Baseline (COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had Haematocrit data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: L/L
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 173 | 178
L/L | 2.8 [2.3 to 3.2] | 2.8 [2.3 to 3.2]

23. Secondary Outcome: MCV Levels
Description: Mean Corpuscular volume (MCV) levels at COVID-19 diagnosis
Time Frame: Baseline(COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had MCV data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: fL
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 176 | 181
fL | 91.4 [90.3 to 92.5] | 87.3 [86.0 to 88.6]

24. Secondary Outcome: MCH Levels
Description: Mean Corpuscular Haemoglobin levels at COVID-19 diagnosis
Time Frame: Baseline(COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had MCH data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: pg
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 171 | 175
pg | 30.2 [29.8 to 30.7] | 29.1 [28.7 to 29.4]

25. Secondary Outcome: HbA1C Levels
Description: Glycated Haemoglobin (HbA1C) levels at COVID-19 diagnosis
Time Frame: Baseline(COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had HbA1C data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mmol/mol
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 4 | 4
mmol/mol | 60.5 [2.1 to 118.9] | 99.2 [15.4 to 213.7]

26. Secondary Outcome: C-reactive Protein Levels
Description: C-reactive protein levels at COVID-19 diagnosis
Time Frame: Baseline(COVID-19 diagnosis)
Population: The analyses was performed with PLHIV with COVID-19 and matched HIV-uninfected with COVID-19 patients. The endpoint is only applicable to patients with COVID-19, therefore data is not reported for the PLWHIV without COVID-19 group. Due to the retrospective nature of this data collection study, not all patients in the PLWHIV+COVID-19+ and the HIV-COVID-19 + groups had CRP data available and could not be included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
Number analyzed (Participants) | 129 | 131
mg/L | 12.6 [9.3 to 15.8] | 13.6 [9.9 to 17.4]

27. Primary Outcome: Time Since HIV Diagnosis
Description: Identification of risk factors for COVID-19 infection within the group of PLHIV: Time since HIV diagnosis
Time Frame: Baseline(Last CD4 cell count and HIV-RNA before COVID-19 diagnosis, or most recent for PLHIV without COVID-19)
Population: as for outcome 6
Measure: Number; unit: per 10 unit of the model
Arm/Group | PLWHIV With COVID-19 Cases | PLWHIV Without COVID-19 Controls
Number analyzed (Participants) | 500 | 992
per 10 unit of the model | 17.1 | 18.3
Statistical Analysis 1: Comparison: PLWHIV With COVID-19 Cases vs PLWHIV Without COVID-19 Controls; Conditional logistic regression models accounting for case-control matching will be used to identify risk factors for advanced immunodeficiency associated with COVID-19. Odds ratio (OR), and the 95% confidence intervals of the OR will be calculated; Test type: Other; p = 0.033, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.74 to 0.99]

28. Primary Outcome: Chronic Obstructive Pulmonary Disease
Description: Identification of risk factors for COVID-19 infection within the group of PLHIV: Chronic Obstructive Pulmonary Disease
Time Frame: Baseline(Last CD4 cell count and HIV-RNA before COVID-19 diagnosis, or most recent for PLHIV without COVID-19)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | PLWHIV With COVID-19 Cases | PLWHIV Without COVID-19 Controls
Number analyzed (Participants) | 500 | 992
participants | 36 | 43
Statistical Analysis 1: Comparison: PLWHIV With COVID-19 Cases vs PLWHIV Without COVID-19 Controls; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.16 to 3.22]

29. Primary Outcome: CD4 Cell Count
Description: Identification of risk factors for COVID-19 infection within the group of PLHIV: CD4 cell count
Time Frame: Baseline(Last CD4 cell count and HIV-RNA before COVID-19 diagnosis, or most recent for PLHIV without COVID-19)
Population: as for outcome 6
Measure: Number; unit: per 100 unit for the model
Arm/Group | PLWHIV With COVID-19 Cases | PLWHIV Without COVID-19 Controls
Number analyzed (Participants) | 500 | 992
per 100 unit for the model | 630 | 630
Statistical Analysis 1: Comparison: PLWHIV With COVID-19 Cases vs PLWHIV Without COVID-19 Controls; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.458, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.95 to 1.02]

30. Primary Outcome: Chronic Kidney Disease
Description: Identification of risk factors for COVID-19 infection within the group of PLHIV: Chronic Kidney Disease
Time Frame: Baseline(Last CD4 cell count and HIV-RNA before COVID-19 diagnosis, or most recent for PLHIV without COVID-19)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | PLWHIV With COVID-19 Cases | PLWHIV Without COVID-19 Controls
Number analyzed (Participants) | 500 | 992
participants | 38 | 32
Statistical Analysis 1: Comparison: PLWHIV With COVID-19 Cases vs PLWHIV Without COVID-19 Controls; [analysis description as in outcome 27, analysis 1]; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.61 to 4.57]

31. Primary Outcome: Body Weight
Description: Identification of risk factors for COVID-19 infection within the group of PLHIV: Body weight
Time Frame: Baseline(Last CD4 cell count and HIV-RNA before COVID-19 diagnosis, or most recent for PLHIV without COVID-19)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | PLWHIV With COVID-19 Cases | PLWHIV Without COVID-19 Controls
Number analyzed (Participants) | 500 | 992
kg | 80 [70 to 91] | 77 [68 to 88]
Statistical Analysis 1: Comparison: PLWHIV With COVID-19 Cases vs PLWHIV Without COVID-19 Controls; [analysis description as in outcome 27, analysis 1]; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.34 to 2.25]

ADVERSE EVENTS:
Time Frame: Baseline to week 6
Description: Adverse events were not assessed were for this study, only deaths and serious adverse events were recorded(hospitalisations).
Arm/Group | PLWHIV With COVID-19 Cases | HIV Seronegative Patients With COVID-19 Controls
All-Cause Mortality (participants affected / at risk) | 24/486 | 23/1106
Serious Adverse Events (participants affected / at risk) | 224/486 | 231/1106
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLWHIV With COVID-19 Cases (N=486) | HIV Seronegative Patients With COVID-19 Controls (N=1106)
Mortality (General disorders) | 24 | 23 — All cause mortality
Hospitalisation (General disorders) | 200 | 208 — In patient hospitalisation

LIMITATIONS AND CAVEATS:
There are two analysis groups: exposed/unexposed (HIV+COVID-19+ and HIV-COVID-19+) and case-control (HIV+COVID-19+ and HIV+COVID-19-). There are limitations in data availability as this is a retrospective data collection study and all variables could not be collected for all participants. Multiple imputation using Chained Equations approach (MICE) was used to fill in missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT05481216/Prot_SAP_000.pdf